CLINICAL TRIAL: NCT00762112
Title: A Long-Term, Open-Label, Phase 3a Safety Study of Oral TAK-559 (32 mg QD) in the Treatment of Patients With Type 2 Diabetes Mellitus
Brief Title: Safety Study of TAK-559 in Treating Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Hepatic safety signal identified.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-03-TL-559-017; U1111-1128-4850 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy.
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — (E)-4-(4-((5-methyl-2-phenyl-1,3-oxazol-4-yl)methoxy)benzyloxyimino)-4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-559 32 mg QD (Experimental)
  Interventions: Drug: TAK-559

INTERVENTIONS:
Drug: TAK-559 — TAK-559 32 mg, tablets, orally, once daily for up to 24 months.

SUMMARY:
The purpose of this study was to determine the long-term safety of TAK-559, once daily (QD), in subjects with Type 2 Diabetes.

DETAILED DESCRIPTION:
Insulin is a primary regulator of blood glucose concentrations. A subnormal response to circulating insulin levels at target tissues leads to a decrease in insulin-mediated glucose uptake. Insulin resistance is associated with normal to high insulin levels and is often accompanied by dyslipidemia, a disruption in lipid metabolism resulting in increased triglycerides and low-density lipoprotein levels as well as decreased high-density lipoprotein levels in patients with type 2 diabetes mellitus. In the early stages of insulin resistance, a compensatory mechanism of increased insulin secretion by the pancreas maintains normal to near-normal glucose levels. Once the pancreas fails to maintain the increased insulin output, overt type 2 diabetes mellitus occurs.

Insulin also plays an important role in the metabolism of fat and proteins and exerts its influence at the peroxisome proliferator-activated receptor level. Peroxisome proliferator-activated receptor -alpha receptors are expressed predominantly in skeletal muscle, adipose tissue, heart, liver, kidney, gut, macrophages, and vascular tissue, and play a key role in energy storage, glucose homeostasis, and vascular biology. Thus, as insulin activates peroxisome proliferator-activated receptor-alpha receptors, this results in the cellular uptake of glucose. Peroxisome proliferator-activated receptor receptors are ligand-activated transcription elements that regulate gene expression necessary for metabolism. For this reason, peroxisome proliferator-activated receptors play a pivotal role in glucose homeostasis, adipocyte differentiation, and lipid storage. The genes predominantly targeted by transcription activity of activated peroxisome proliferator-activated receptor-alpha receptors are those that mediate fatty acid uptake, fatty acid oxidation, and lipoprotein metabolism. As such, peroxisome proliferator-activated receptor-alpha agonists have their greatest effect on lipid metabolism and vascular biology.

TAK-559 is a novel oxyiminoalkanoic acid under investigation for use as an oral agent in the treatment of patients with type 2 diabetes mellitus. TAK-559 has partial peroxisome proliferator-activated receptor-alpha agonist activity, potent peroxisome proliferator-activated receptor-alpha activity, and modest peroxisome proliferator-activated receptor-gamma activity at high concentrations in nonclinical models.

ELIGIBILITY:
Inclusion Criteria:

* Required sponsor approval if older than 80 years.
* Had either:

  * Successfully completed Protocol 01-03-TL-559-016, or
  * Participated in either Protocol 01-02-TL-559-013, 01-02-TL-559-014, 01-04-TL-559-028, or 01-04-TL-559-029 and either

    * completed the study
    * prematurely terminated from the study due to the HbA1c withdrawal criterion after at least 12 weeks of treatment, or
    * in the opinion of the investigator, demonstrated a lack of efficacy after at least 16 weeks of treatment and was withdrawn from the study.
* A female subject of childbearing potential who was sexually active agreed to use adequate contraception, and was neither pregnant nor lactating from Screening throughout the duration of the study.
* Were willing to continue following an individualized weight maintenance diet during the study period.
* Had evidence of insulin secretory capacity, as demonstrated by a fasting C-peptide concentration of greater than or equal to 1.5 ng/mL (0.50 nmol/L) at the prior visit of Protocol 013, 014, 016, 028, or 029.
* Were willing to perform daily self-monitoring blood glucose tests.
* Were in good health at Enrollment, as determined by a physician at the final visit of Protocol 013, 014, 016, 028, or 029 (ie, via medical history and physical examination), other than having type 2 diabetes mellitus and New York Heart Association Classification I or II congestive heart failure.
* Had clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis after fasting for at least 8 hours) within the normal reference range for the testing laboratory, unless the results were deemed not clinically significant by the investigator or sponsor, at the prior visit of Protocol 013, 014, 016, 028, or 029.
* Had a normal thyroid-stimulating hormone level of less than 5.5 uIU/mL (5.5 mIU/L) and greater than or equal to 0.35 uIU/mL (0.35 mIU/L) at the prior visit of Protocol 013, 014, 016, 028, or 029.

Exclusion Criteria:

* Had significant cardiovascular disease, including, but not limited to, New York Heart Association Classification III or IV CHF at Enrollment.
* Had a planned surgical or catheter intervention for coronary angioplasty within 12 months after the Enrollment Visit.
* Had a systolic blood pressure greater than 140 mm Hg or a diastolic blood pressure greater than 95 mm Hg at Enrollment.
* Had symptomatic orthostatic hypotension or systolic blood pressure less than 90 mm Hg at Enrollment.
* Had a history of a clinically significant abnormal electrocardiogram or experienced any cardiovascular event including, but not limited to, myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, or documented cerebrovascular accident during Protocol 013, 014, 016, 028, or 029.
* Had a creatine phosphokinase value above 3 times the upper limit of normal at the prior visit of Protocol 013, 014, 016, 028, or 029.
* Had a triglyceride level greater than 500 mg/dL (5.6 nmol/L) at the prior visit of Protocol 013, 014, 016, 028, or 029.
* Had an alanine aminotransferase or aspartate aminotransferase level above 3 times the upper limit of normal, active liver disease, or jaundice at any time during Protocol 013, 014, 016, 028, or 029.
* Had donated and/or received any blood products within 3 months prior to Enrollment.
* Had used illicit drugs or abused alcohol during participation in Protocol 013, 014, 016, 028, or 029.
* Had experienced another illness occurring at the same time requiring hospitalization during the occurring at the same time 3 weeks before the Enrollment Visit.
* Had experienced any other serious disease or condition during participation in Protocol 013, 014, 016, 028, or 029 that might have affected life expectancy or made it difficult to successfully manage and follow the patient according to the protocol.
* Was required to take or intended to continue taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfered with the evaluation of the study medication, including:

  * insulin (for patients who participated in Protocol 01-02-TL-559-013, 01-02-TL-559-014, 01-04-TL-559-028, and 01-04-TL-559-029)
  * prescription-strength niacin
  * fibric acid derivatives
  * systemic corticosteroids
  * warfarin
  * rifampin
  * nicotinic acid
  * St. John's Wort
  * thiazolidinediones
  * peroxisome proliferator-activated receptor agonists other than the study drug.
* Had experienced persistent unexplained microscopic or macroscopic hematuria or developed cancer of the bladder while participating in Protocol 013, 014, 016, 028, or 029.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2003-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinical laboratory hematology tests. | Week 2 and Months 6, 12, 18, and Final Visit
Change from baseline in clinical laboratory chemistry tests. | Week 2 and Months 6, 12, 18, and Final Visit
Blood pressure measurements. | All visits.
Pulse measurements. | All visits.
Body weight. | All visits.
Physical examinations. | Months 6, 12, 18, and Final Visit
12-lead electrocardiogram. | Months 6, 12, and Final Visit
Adverse event occurrence. | All visits or at occurrence

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Months 3, 6, 9, 12, 15, 18, 21, and Final Visit
Change from baseline in fasting plasma glucose. | All visits.
Change from baseline in fasting insulin. | Months 3, 6, 9, 12, 15, 18, 21, and Final Visit
Change from baseline in fasting C-peptide. | Months 6, 12, 18, and Final Visit
Change from baseline in triglycerides. | Months 6, 12, 18, and Final Visit
Change from baseline in total cholesterol. | Months 6, 12, 18, and Final Visit
Change from baseline in high-density lipoprotein. | Months 6, 12, 18, and Final Visit
Change from baseline in low-density lipoprotein. | Months 6, 12, 18, and Final Visit
Change from baseline in very-low-density lipoprotein. | Months 6, 12, 18, and Final Visit
Change from baseline in low-density lipoprotein fractionation. | Months 6, 12, 18, and Final Visit
Change from baseline in intermediate-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in large low-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in small low-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in medium-small low-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in very-small low-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in mean low-density lipoprotein size. | Months 6, 12, 18, and Final Visit
Change from baseline in apolipoproteins A1 and B. | Months 12 and Final Visit
Change from baseline in atherosclerosis marker plasminogen activator inhibitor 1. | Months 6, 12, and Final Visit
Change from baseline in atherosclerosis marker fibrinogen. | Months 6, 12, and Final Visit
Change from baseline in inflammation marker Interleukin-6. | Months 6, 12, and Final Visit
Change from baseline in inflammation marker C-reactive protein. | Months 6, 12, and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda